CLINICAL TRIAL: NCT02174614
Title: The Effect of Cognitive Enhancement as a Precursor to Computer Based Training for Cognitive Behavioral Therapy (CBT4CBT)
Acronym: Project 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1405013937; 2P50DA009241-21 (NIH)
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Cocaine Use Disorder
Keywords: Cocaine use disorder
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment As Usual (TAU) (Active Comparator): Treatment normally offered at this clinic which could include individual or group drug counseling sessions three times per week lasting three hours each time.
  Interventions: Behavioral: Treatment As Usual (TAU)
- TAU plus Rapid Abstinence Initiation (RAI) (Experimental): Treatment normally offered at this clinic which could include individual or group drug counseling sessions three times per week lasting three hours each time PLUS the chance to earn money for urine specimens that are negative for cocaine during the first 4 weeks of treatment
  Interventions: Behavioral: Treatment As Usual (TAU); Behavioral: TAU plus Rapid Abstinence Initiation (RAI)
- TAU plus RAI plus Cognitive Control Training (CCT) (Experimental): Treatment normally offered at this clinic which could include individual or group drug counseling sessions three times per week lasting three hours each time PLUS the chance to earn money for urine specimens that are negative for cocaine during the first 4 weeks of treatment PLUS sessions of computerized games 3 times per week for the first 4 weeks.
  Interventions: Behavioral: Treatment As Usual (TAU); Behavioral: TAU plus Rapid Abstinence Initiation (RAI); Behavioral: TAU plus RAI plus Cognitive Control Training (CCT)

INTERVENTIONS:
Behavioral: Treatment As Usual (TAU) — Treatment normally offered at this clinic which could include individual or group drug counseling sessions three times per week lasting three hours each time.
Behavioral: TAU plus Rapid Abstinence Initiation (RAI) — Treatment normally offered at this clinic which could include individual or group drug counseling sessions three times per week lasting three hours each time PLUS the chance to earn money for urine specimens that are negative for cocaine during the first 4 weeks of treatment followed by 8 weeks of CBT4CBT computerized therapy.
  Arms: TAU plus RAI plus Cognitive Control Training (CCT); TAU plus Rapid Abstinence Initiation (RAI)
Behavioral: TAU plus RAI plus Cognitive Control Training (CCT) — Treatment normally offered at this clinic which could include individual or group drug counseling sessions three times per week lasting three hours each time PLUS the chance to earn money for urine specimens that are negative for cocaine during the first 4 weeks of treatment PLUS sessions of computerized cognitive control training (CCT) 3 times per week for the first 4 weeks followed by 8 weeks of CBT4CBT computerized therapy.
  Arms: TAU plus RAI plus Cognitive Control Training (CCT)

SUMMARY:
The investigators are conducting a randomized clinical trial of rapid abstinence initiation and cognitive control training as a precursor to our new web-based version of the CBT4CBT (Computer Based Training for Cognitive Behavioral Therapy) program to evaluate its effectiveness relative to standard outpatient counseling at the Midwestern Connecticut Council of Alcoholism (MCCA). CCT will be used to assess attention, working memory and inhibitory control and the computer-based training program (CBT4CBT) focuses on teaching basic coping skills, presenting examples of effective use of coping skills in a number of realistic situations in video form, and providing opportunities for patients to practice and review new skills while receiving cocaine abuse treatment.

DETAILED DESCRIPTION:
150 cocaine dependent individuals will be randomly assigned to one of 3 conditions delivered over 4 weeks in the context of intensive outpatient treatment. 1. Treatment as Usual (TAU), 2. rapid abstinence initiation (RAI) or 3. computerized cognitive control training with escalating reinforcement for improved performance on training tasks (CCT). All participants will then receive an 8 week trial of CBT4CBT in addition to TAU. Follow up evaluation thru 6 months posttreatment will assess durability and delayed emergence of treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Meet current DSM-5 criteria for cocaine use disorder
* Are sufficiently stable for 12 weeks of outpatient treatment
* Are willing to provide locator information for follow-up
* Are fluent in English
* Have a 6th grade or higher reading level for completion of assessments

Exclusion Criteria:

* Untreated bipolar or schizophrenic disorder
* Current suicide risk
* Have a legal case pending such that incarceration during the 12-week protocol is likely
* Are physically dependent on alcohol, opioids or benzodiazepines and require detoxification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Reduction in cocaine use | 12 weeks
  Using urine and breathalyzer screening for negative cocaine and alcohol testing.

SECONDARY OUTCOMES:
Subjects ability to demonstrate coping skills acquisition through a computerized role-playing evaluation | 12 weeks
  Use of CBT4CBT program with acquisition of skills demonstrated through homework assignments.

OTHER OUTCOMES:
Increased cognitive function and working memory | 12 weeks
  development of skills used in attention, working memory and inhibitory control as demonstrated through an extensive assessment battery.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kiluk, PhD, Study Director — Yale University
Locations (2):
- United States (2):
  - MCCA, Bridgeport, Connecticut
  - MCCA, New Haven, Connecticut